CLINICAL TRIAL: NCT04177277
Title: Dialysis mHealth Survey (mHealth Access and Usage by Dialysis Patients and Staff)
Brief Title: Dialysis mHealth Survey
Status: Completed | Type: Observational
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: SIH119_mHealth
Record Dates: First submitted 2019-11-20; First posted 2019-11-26 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: ESRD
Keywords: Dialysis; mHealth
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a survey of dialysis patients and staff to determine both the readiness of ESRD patients to use mHealth as well as the Readiness of the dialysis center staff (healthcare technicians, nurses and administrative staff) to utilize mHealth in order to assist patients who may have barriers to do so for themselves.

DETAILED DESCRIPTION:
This is a cross-sectional observational study. Approximately 700 ESRD patients currently on dialysis will be recruited from Satellite In-Center (Hemodialysis) and WellBound (Home Dialysis) Centers in the US. These will include centers in Texas, Tennessee, and California. In addition, about 100 dialysis staff will be recruited to complete a staff mHealth Questionnaire.

Patients and staff will be asked questions that conform to Khatun's conceptual model.

* Technological readiness:

  * Availability of the devices and internet
  * Ability to use the devices
* Human resource readiness:

  * Socio-demographics
  * Awareness of mHealth services
* Motivational readiness

  * Concerns (cost/privacy/ other)
  * Attitudes/intentions: Current use or potential for use.

ELIGIBILITY:
Inclusion Criteria:

* • On dialysis (either in-center or home) at a participating Satellite Healthcare center within the recruitment period

  * Any Satellite Dialysis staff member with patient interaction.

Exclusion Criteria:

* Age < 18 years
* Inability to participate because of cognitive impairment or active psychological condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Dialysis patients and staff at participating centers (both in-center and home-based) who volunteer to participate in the study by completing the one-time survey. Centers selected for participation were in California, Tennessee, and Texas.
Sampling Method: Non-Probability Sample
Enrollment: 949 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who have access to and ability to use smart devices and the internet | One day
  Number of Patients who have access compared to all patients surveyed
Percentage of patients aware of mHealth Services | One day
  Number of patients who have awareness of websites, apps or other sites used for self mobile health compared to al patients surveyed
Common Concerns of patients regarding mHealth | One day
  Survey question regarding potential concerns in usage of self mobile health resources
Percentage of patients who currently use or would use mHealth services | One day
  Number of patients who use MHealth compared to all patients surveyed
Relationship of Age to mHealth usage | One day
  statistical analysis
Relationship of Gender to mHealth usage | One day
  statistical analysis
Relationship of Ethnicity to mHealth usage | one day
  statistical analysis
Relationship of Insurance Coverage to mHealth usage | one day
  statistical analysis
Relationship of Employment to mHealth usage | one day
  statistical analysis

SECONDARY OUTCOMES:
Percentage of staff who have access and ability to use smart devices and the internet | One day
  Number of staff who have access compared to all patients surveyed
Percentage of staff who would be comfortable assisting patients to utilize mHealth Services | One day
  Number of staff comfortable compared to all staff surveyed
Relationship of Staff age to smart device use and willingness to assist | One day
  Analysis
Relationship of Staff position to smart device use and willingness to assist | One day
  Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Wael F Hussein, MBBS, Principal Investigator — Satellite Healthcare, Inc.
Locations (1):
- Satellite Healthcare, Inc., San Jose, California, United States

REFERENCES:
- [Derived] Hussein WF, Bennett PN, Pace S, Chen S, Legg V, Atwal J, Sun S, Schiller B. The Mobile Health Readiness of People Receiving In-Center Hemodialysis and Home Dialysis. Clin J Am Soc Nephrol. 2020 Dec 31;16(1):98-106. doi: 10.2215/CJN.11690720. Epub 2020 Dec 22. PMID 33355235